CLINICAL TRIAL: NCT05410795
Title: Establishment and Verification of Pancreatic Volume Formula Based on Imaging: A Cross-sectional Study
Brief Title: Establishment and Verification of Pancreatic Volume Formula Based on Imaging
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: EPIC20220428
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy People; Chronic Pancreatitis; Acute Pancreatitis
Keywords: Magnetic resonance imaging; Pancreatic volume
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy people: Healthy people refer to those who exclude pancreatic related diseases, such as acute and chronic pancreatitis, pancreatic trauma, pancreatic tumor, peripancreatic lesions, diabetes and other diseases that may affect the volume of the pancreas.
  Interventions: Diagnostic Test: Magnetic resonance imaging
- Chronic pancreatitis: Patients with chronic pancreatitis are considered as study subjects.
  Interventions: Diagnostic Test: Magnetic resonance imaging
- Acute pancreatitis: Patients with acute pancreatitis within 144 hours after the onset of typical symptoms are considered as study subjects.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Enrolled subjects will be examined with MRI of pancreas, and the volume, length and thickness of coronal plane of pancreas will be measured by software.

SUMMARY:
This study intends to construct the linear relationship between pancreatic volume and individual attributes (height, weight, width of anterior superior iliac spine, etc.), and to establish and verify the formula of pancreatic volume.

DETAILED DESCRIPTION:
The volume of pancreas in healthy individuals changes with age. The pancreatic volume gradually increases from birth to 20 years old. There is a plateau period from 20 to 60 years old, and the volume gradually decreases after 60 years old. With the development of imaging technology, pancreatic volume can be measured by computer tomography and magnetic resonance imaging.

Whether it is pancreatic atrophy after chronic pancreatitis or pancreatic edema after acute pancreatitis, the pathological changes of pancreatic parenchyma may lead to changes in pancreatic volume. Many studies have confirmed that pancreatic volume can be used to evaluate the course of pancreatic related diseases such as diabetes and acute pancreatitis.

Therefore, the establishment of accurate and convenient pancreatic volume formula can help to estimate the initial pancreatic volume of patients. This study is helpful to evaluate the clinical stage, severity and prognosis of pancreatic related diseases.

ELIGIBILITY:
Inclusion Criteria (Meet 1 or 2 or 3):

* Healthy individuals (excluding pancreatic related diseases, such as acute and chronic pancreatitis, pancreatic trauma, pancreatic tumor, peripancreatic lesions, diabetes and other diseases that may affect the volume of the pancreas);
* Patients with chronic pancreatitis;
* Patients with acute pancreatitis within 144 hours after the onset of typical symptoms (severe persistent epigastric pain).

Exclusion Criteria:

* suspected to have malignant tumors;
* History of pancreas related surgery or minimally invasive treatment (such as pancreaticoduodenectomy, ERCP, etc.);
* acute exacerbation of chronic pancreatitis;
* pregnant or breastfeeding women;
* patients who refused to participate in the study.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients meeting the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pancreatic volume | 14 days after MRI examination
  The total volume of pancreas and the volumes of head, body and tail of pancreas will be calculated by software.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No